CLINICAL TRIAL: NCT06540482
Title: Reliability and Validity of the Figure of 8 Walk Test With and Without Dual-Task in Individuals With Stroke
Brief Title: Reliability and Validity of The Figure of 8 Walk Test With and Without Dual-Task
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Associate Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 07.05.2022-09
Record Dates: First submitted 2024-07-31; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Stroke
Keywords: stroke; validity and reliability
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke patients: The participants consisted of stroke patients aged 50 years and older who were followed up and treated by Pamukkale University Adult Neurological Rehabilitation - Outpatient Unit.
  Interventions: Diagnostic Test: Reliability test

INTERVENTIONS:
Diagnostic Test: Reliability test — The test was administered two days apart to evaluate the reliability of the retest test.

SUMMARY:
For people with stroke, walking on a curved path is more difficult than walking on a straight path and can lead to falls. Most of the outcome scales assessing the gait of people with stroke involve walking in a straight line or with one turn. Assessing a person with stroke walking on a straight path may not be indicative of real-life gait-related performance. The Figure of 8 Walk Test (F8WT) includes a straight and curved gait that may represent the daily gait. To the best of our knowledge, there are no studies evaluating the reliability and validity of the dual-task F8W test in individuals with stroke. Therefore, the aim of this study was to evaluate the validity and reliability of the F8W and dual-task F8W test in individuals with stroke.

DETAILED DESCRIPTION:
For people with stroke, walking on a curved path is more difficult than walking on a straight path and can lead to falls. Most of the outcome scales assessing the gait of people with stroke involve walking in a straight line or with one turn. Assessing a person with stroke walking on a straight path may not be indicative of real-life gait-related performance. The Figure of 8 Walk Test (F8WT) includes a straight and curved gait that may represent the daily gait. To the best of our knowledge, there are no studies evaluating the reliability and validity of the dual-task F8W test in individuals with stroke. Therefore, the aim of this study was to evaluate the validity and reliability of the F8W and dual-task F8W test in individuals with stroke.

This prospectively designed study evaluated the demographic and clinical characteristics of the participants. The main outcome measures included the F8WT, dual-task F8WT, Standardised Mini Mental Test, The National Institutes of Health Stroke Scale, Timed-Up and Go Test, 10-metre walk test, Modified Four Square Step Test and Six-Spot Step Test.

ELIGIBILITY:
Inclusion Criteria:

* 50 years of age or older,
* Having had only one unilateral stroke at least 6 months before the study,
* Being medically stable,
* Being able to walk at least 10 metres with a cane or independently,
* Getting at least 24 points from the Standardised Mini Mental Test,
* Being able to perform the cognitive task (subtraction) given during the assessments.

Exclusion Criteria:

* Presence of additional orthopaedic, neurological or cardiovascular diseases that may affect balance and walking,
* Uncorrectable visual and hearing problems

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants consisted of stroke patients aged 50 years and older who were followed up and treated by Pamukkale University Adult Neurological Rehabilitation-Outpatient Unit
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-09-25 (Actual); Primary Completion 2024-07-25 (Actual); Study Completion 2024-07-25 (Actual)

PRIMARY OUTCOMES:
The Figure of 8 Walk Test (F8WT) | The test will be administered first and third day.
  The test starts from the center of two cones at a certain distance. Participants are asked to walk around the cones in 8 shapes at their normal walking speed. The test ends when the participant reaches the starting point again. The duration of the test is recorded in seconds.
Dual-task The Figure of 8 Walk Test (F8WT) | The test will be administered first and third day.
  The test starts from the center of two cones at a certain distance. Participants were asked to walk around the cones in 8 shapes at their normal walking speed when they conducted the cognitive or motor task. The test ends when the participant reaches the starting point again. The duration of the test is recorded in seconds.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No